CLINICAL TRIAL: NCT03011996
Title: An Open-label, Randomized Study to Evaluate Pharmacokinetic Interaction, Pharmacodynamics and Safety After Multiple Oral Dosing of CJ-12420 and Amoxicillin/Clarithromycin in Healthy Subjects
Brief Title: To Investigate PK and PD of CJ-12420, Clarithromycin, Amoxicillin After Multiple Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_APA_107
Record Dates: First submitted 2016-12-13; First posted 2017-01-06 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Drug Interaction; Pharmacokinetic; Pharmacodynamic
MeSH Terms: interventions — Clarithromycin; Amoxicillin; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- CJ-12420 100mg (Experimental): CJ-12420 100mg BID for 5 days
  Interventions: Drug: CJ-12420 100mg
- CJ-12420 50mg + CLR 500mg + AMX 1g (Experimental): coadministration of CJ-12420 50mg and CLR 500mg/AMX 1g BID for 7 days
  Interventions: Drug: CLR 500mg; Drug: CJ-12420 50mg; Drug: AMX 1g
- Pantoprazole 40mg + CLR 500mg + AMX 1g (Active Comparator): coadministration of Pantoprazole 40mg and CLR 500mg/AMX 1g BID for 7 days
  Interventions: Drug: CLR 500mg; Drug: AMX 1g; Drug: Pantoprazole 40mg
- CJ-12420 100mg + CLR 500mg + AMX 1g (Experimental): coadministration of CJ-12420 100mg, CLR 500mg/AMX 1g BID for 7 days
  Interventions: Drug: CLR 500mg; Drug: CJ-12420 100mg; Drug: AMX 1g
- CLR 500mg/AMX 1g (Experimental): CLR 500mg/AMX 1g BID for 5 days
  Interventions: Drug: CLR 500mg; Drug: AMX 1g
- CJ-12420 100mg + CLR 500mg/AMX 1g (Experimental): coadministration of CJ-12420 100mg and CLR 500mg/AMX 1g BID for 7 days
  Interventions: Drug: CLR 500mg; Drug: CJ-12420 100mg; Drug: AMX 1g

INTERVENTIONS:
Drug: CLR 500mg — Cohort 1: bid for 5 days Cohort 2: bid for 7 days
  Other Names: Clarithromycin 500mg
  Arms: CJ-12420 100mg + CLR 500mg + AMX 1g; CJ-12420 100mg + CLR 500mg/AMX 1g; CJ-12420 50mg + CLR 500mg + AMX 1g; CLR 500mg/AMX 1g; Pantoprazole 40mg + CLR 500mg + AMX 1g
Drug: CJ-12420 100mg — Cohort 1: bid for 5 days Cohort 2: bid for 7 days
  Arms: CJ-12420 100mg; CJ-12420 100mg + CLR 500mg + AMX 1g; CJ-12420 100mg + CLR 500mg/AMX 1g
Drug: CJ-12420 50mg — Cohort 2: bid for 7 days
  Arms: CJ-12420 50mg + CLR 500mg + AMX 1g
Drug: AMX 1g — Cohort 1: bid for 5 days Cohort 2: bid for 7 days
  Other Names: Amoxicillin 1g
  Arms: CJ-12420 100mg + CLR 500mg + AMX 1g; CJ-12420 100mg + CLR 500mg/AMX 1g; CJ-12420 50mg + CLR 500mg + AMX 1g; CLR 500mg/AMX 1g; Pantoprazole 40mg + CLR 500mg + AMX 1g
Drug: Pantoprazole 40mg — Cohort 2: bid for 7 days
  Arms: Pantoprazole 40mg + CLR 500mg + AMX 1g

SUMMARY:
Cohort 1

To evaluate the pharmacokinetic interactions of CJ-12420 after multiple oral doses of CJ-12420 given alone or in combination with amoxicillin/clarithromycin in healthy subjects.

Cohort 2

To evaluate the pharmacodynamic profiles of CJ-12420 after multiple oral doses of CJ-12420 in combination with amoxicillin/clarithromycin in healthy subjects as compared to an active control group, i.e., pantoprazole in combination with amoxicillin/clarithromycin.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic the drug-drug interaction of CJ-12420 and amoxicillin/clarithromycin and investigate the pharmacodynamic of co-administration of CJ-12420 and amoxicillin and clarithromycin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged ≥19 and ≤45 years at screening;
2. No congenital or chronic disease, and no morbid symptoms or findings on screening tests;
3. Body mass index (BMI) ≥18.5 and ≤28 kg/m2;
4. Considered eligible based on medical examinations (including interview, vital signs, 12-lead ECG, physical exam and laboratory tests) which are set and performed in accordance with the nature of investigational product by the investigator;
5. Voluntary consent to participate in the study after being fully informed of purpose and procedures of the study, and profiles of investigational product prior to the participation;
6. For Cohort 2, positive on 13C urea breath test.

Exclusion Criteria:

1. Medical history

   1. History or current evidence for diseases considered clinically relevant by the investigator including hepatic, renal, gastrointestinal, respiratory, musculoskeletal, endocrine, neurologic, hemato-oncological, urinary, or cardiovascular (including cardiac arrhythmia) diseases;
   2. History of gastrointestinal diseases (such as gastritis, gastrodynia, gastroesophageal reflux disease, Crohn's disease and ulcer) or abdominal surgery (except for simple appendectomy or herniotomy) which are considered to have potential effect on drug absorption by the investigator;
   3. For Cohort 2, previous treatment failure for H. pylori eradication.
2. Laboratory tests and ECG

   1. AST or ALT ≥ 1.25 x upper limit of normal (ULN);
   2. Total bilirubin ≥ 1.5 x ULN;
   3. eGFR calculated by CKD-EPI formula < 80 mL/min;
   4. Any clinically relevant ECG abnormalities.
3. Allergy and drug abuse

   1. History of hypersensitivity to drugs containing investigational products (penicillins, cephems, macrolides, pantoprazole and benzimidazole) and other drugs (including aspirin and antibiotics);
   2. History of drug abuse or positive on drug screening test.
4. Drug/dietary restrictions

   1. Medications (including herbal supplements) or abnormal diet (e.g., grapefruit juice > 1 L/day, excessive garlic, broccoli, kale, etc.) which may have effect on absorption, distribution, metabolism and excretion of investigational products within 28 days prior to the first study dose;
   2. Use of prescription drugs, over-the-counter drugs (OTCs) or vitamins within 10 days prior to the first study dose;
   3. Participating in other study and receive investigational product within 3 months prior to the first study dose.
5. Blood donation and transfusion

   1. Whole blood donation within 60 days prior to the first study dose;
   2. Donation of blood components or transfusion within 30 days prior to the first study dose.
6. Pregnancy and contraception

   1. Pregnant or breast-feeding;
   2. Subject or his partner's inability to use of medically qualifying dual-contraceptive methods or medically acceptable contraception (including intrauterine device with established pregnancy failure rate, barrier methods with spermicide, vasectomy, tubectomy, tubal ligation and hysterectomy) from screening to 30 days of the last dose of investigational product.
7. Others

   1. Heavy use of alcohol (average alcohol intake ≥30 g/day) or positive on alcohol test;
   2. Heavy smoker (>10 cigarettes/day);
   3. Caffeine intake > 400 mg/day;
   4. Any clinically relevant findings considered inappropriate for study participation at the discretion of the investigator.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of CJ-12420, clarithromycin and amoxicillin | Up to 120 hours

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of CJ-12420, clarithromycin and amoxicillin | Up to 120 hours
Time of maximum observed concentraion(tmax) of CJ-12420, clarithromycin and amoxicillin | Up to 120 hours
Half life(t1/2) of CJ-12420, clarithromycin and amoxicillin | Up to 120 hours
Oral clearance at steady state(CLss/F) of CJ-12420, clarithromycin and amoxicillin | Up to 120 hours
Apparent volume of distribution at steady state(Vdss/F) of CJ-12420, clarithromycin and amoxicillin | Up to 120 hours
median pH | Up to 24 hours
  Data from the pH probe monitoring
Time at pH > 3 (%) | Day -1, Day 1, Day 7 up to 24 hours
  the percent of time the pH as data from the pH probe monitoring
Time at pH > 4 (%) | Day -1, Day 1, Day 7 up to 24 hours
  the percent of time the pH as data from the pH probe monitoring
Time at pH > 6 (%) | Day -1, Day 1, Day 7 up to 24 hours
  the percent of time the pH as data from the pH probe monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, Principal Investigator — Inje university college of medicine Busan Paik Hospital
Locations (1):
- Inje University Busan Baik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided